CLINICAL TRIAL: NCT03080246
Title: Effects of Strength Training on Musculoskeletal Overuse Injuries in Female Runners
Acronym: STARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00034222; W81XWH-16-1-0001 (Other: Army Med R & D Command)
Record Dates: First submitted 2016-06-17; First posted 2017-03-15 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2019-12

CONDITIONS: Overuse Injury
MeSH Terms: conditions — Cumulative Trauma Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength Training Group (Active Comparator): This group will begin coming to the Clinical Research Center (near the undergraduate campus of Wake Forest University) for exercise classes 2-3 days per week for about an hour each day. The investigators also have a site on High Point University's campus. The class will consist of a 10-minute warm-up, a 20-minute strength training period, 15-minutes of neuromuscular (balance/coordination) training, and a 15-minute cool down. These regular exercise classes at Wake Forest and High Point University will go on for 9 months, followed by another 9 months of option to continue at facility, plus follow-up via email and 2 group meetings/runs at Fleet Feet (at around months 12 and 15).
  Interventions: Behavioral: Strength Training Exercise
- Running Group (No Intervention): This group will be observed as they follow their usual run-training routine over the course of 18 months. Emails will be sent biweekly for 18 months to update the research team on injury/training status. The group will attend 5 group meetings/runs at Fleet Feet (at around months 1, 3, 6, 12, and 15). After the 18 months, the participants will be offered a free 8-week strength training program at the Clinical Research Center or High Point University.

INTERVENTIONS:
Behavioral: Strength Training Exercise
  Arms: Strength Training Group

SUMMARY:
The purpose of this study is to look at the effect of strength training in preventing overuse injuries in female runners

DETAILED DESCRIPTION:
This randomized clinical trial will compare the effects of 9-months of strength training to a control group on: (1) injury rates in female runners during the 9 month intervention period, and for 9 months after completing the intervention, and (2) on the potential mechanisms of injury including strength, joint and tissue loading, and psychosocial factors.

ELIGIBILITY:
Inclusion Criteria:

* Female civilian runners between 18-60 years old
* Run at least 5 miles per week for the past 6 months
* No overuse injuries in the past 6 months
* Plan to stay in the area for the next year and a half
* Live less than 30 miles from Wake Forest University or High Point University

Exclusion Criteria:

* Male
* Under age 18 and over age 60
* Chronic diseases, orthopedic conditions, past anterior cruciate ligament tears
* Currently pregnant or planning to conceive within the next 18 months
* Observed by study staff as unwilling to attend testing/intervention sessions
* Observed by study staff as unwilling to communicate via telephone and email regularly with study personnel
* Participated in formal strength training in the past 6 months
* Current active military or active military reserve

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2015-12; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Overuse Injury (Physical Exam/Injury Report Form) | Month 18
  To compare the effects of a 9-month strength training program to a control group on the incidence of overuse, lower extremity, running injuries in female adult recreational and competitive runners during and 9 months subsequent to the training period.

SECONDARY OUTCOMES:
Lower Extremity Muscular Strength (HUMAC norm isokinetic dynamometer) | Months 0, 9, and 18
  To compare the effects of 9-months of strength training to a control group on lower extremity muscular strength at the conclusion and 9 months subsequent to completion of the intervention.
Biomechanical Joint Moments (3D kinematic and kinetic data collected by 6-camera motion capture gait analysis) | Month 0, 9, and 18
  To compare the effects of 9-months of strength training to a control group on hip, knee, and ankle joint moments during running at the conclusion and 9 months subsequent to completion of the intervention.
Biomechanical Joint Forces (3D kinematic and kinetic data collected by 6-camera motion capture gait analysis) | Month 0, 9, and 18
  To compare the effects of 9-months of strength training to a control group on knee and ankle compressive and shear bone-on-bone joint forces during running at the conclusion and 9 months subsequent to completion of the intervention.
Biomechanical Joint Tissue Loading (3D kinematic and kinetic data collected by 6-camera motion capture gait analysis) | Month 0, 9, and 18
  To compare the effects of 9-months of strength training to a control group on joint tissue loading during running at the conclusion and 9 months subsequent to completion of the intervention.
Self-Efficacy (Adherence Self-Efficacy Questionnaire) | Months 0, 9, and 18
  To compare the effects of 9-months of strength training to a control group on performance self-efficacy at the conclusion and 9 months subsequent to completion of the intervention
Quality of Life (SF-12 Health Related Quality of Life Survey) | Months 0, 9, and 18
  To compare the effects of 9-months of strength training to a control group on health-related quality of life at the conclusion and 9 months subsequent to completion of the intervention
Quality of Life (Satisfaction with Life Scale) | Months 0, 9, and 18
  To compare the effects of 9-months of strength training to a control group on health-related quality of life at the conclusion and 9 months subsequent to completion of the intervention
Quality of Life (Positive and Negative Affect Scale) | Months 0, 9, and 18
  To compare the effects of 9-months of strength training to a control group on health-related quality of life at the conclusion and 9 months subsequent to completion of the intervention
Quality of Life (State Trait Anxiety Inventory-S Scale) | Months 0, 9, and 18
  To compare the effects of 9-months of strength training to a control group on health-related quality of life at the conclusion and 9 months subsequent to completion of the intervention
Quality of Life (Visual Analog Pain Scale) | Months 0, 9, and 18
  To compare the effects of 9-months of strength training to a control group on health-related quality of life at the conclusion and 9 months subsequent to completion of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Messier, PhD, Principal Investigator — Wake Forest University
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT03080246/ICF_000.pdf